CLINICAL TRIAL: NCT05614050
Title: The Prognosis of Patients After Coronary Intervention (PCI) : a Multi-center Prospective Study in China
Brief Title: The Prognosis of Patients After PCI：a Multi-center Study in China
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Shandong Provincial Hospital (Other Government); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Xiamen University (Other); Shanxi Cardiovascular Hospital (Other); First People's Hospital of Xianyang (Other); Yichang Central People's Hospital (Other); Jingzhou Central Hospital (Other); The First Hospital of Wuhan (Unknown); Wuhan Central Hospital (Other); Wuhan Fourth Hospital (Unknown); Fifth Hospital in Wuhan (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Wuhan Asia Heart Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Central Hospital of Enshi Tujia and Miao Autonomous Prefecture (Unknown); Hubei University of Medicine (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Director of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: ChiPCI
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and whole blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary artery disease (CAD) is caused by myocardial ischemia, hypoxia or necrosis due to coronary artery stenosis, spasm or obstruction. Although standard drug therapy can greatly improve the prognosis of patients with CAD after percutaneous coronary interventions (PCI), these patients are still at high risk of major adverse cardiovascular and cerebrovascular events (MACCE). At present, the concept of residual inflammation risk (RIR) has aroused widespread concern. RIR is an important independent risk in patients with CAD. Previous studies indicated that hsCRP ≥ 2mg / L was the definition standard of RIR in CAD in European and American people. In China, the impact of dynamic changes of hsCRP and other inflammatory factors on MACCE in PCI population remains unclear. Therefore, in this study, the investigators plan to recruit patients undergoing PCI, and observe the impact of hsCRP and other inflammatory factors on the prognosis of these patients during long term follow-up at 17 hospitals in China.

ELIGIBILITY:
Inclusion Criteria:

* Participants who understand and sign the informed consent voluntarily;
* Age ≥ 18 years old and ≤ 80 years old, regardless of sex;
* The hospitalized patients with coronary heart disease undergoing PCI;
* Complete all planned PCI during hospitalization.

Exclusion Criteria:

* Acute, chronic or recurrent infectious diseases;
* Immune diseases or immune-related diseases;
* Long-term use of non-steroidal anti-inflammatory drugs, hormones, immunomodulatory and chemotherapy drugs;
* Pregnant women, lactating women or women of childbearing age who do not use effective contraceptive measures;
* The researchers determined that other conditions in which the patient was not suitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The hospitalized patients with coronary heart disease completing all planned PCI
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
MACCE | 12 months
  A composite of all-cause death, nonfatal myocardial infarction, nonfatal stroke, ischemia-driven revascularization

SECONDARY OUTCOMES:
all-cause death | 12 months
  Occurrence of all-cause death
cardiovascular death | 12 months
  Occurrence of cardiovascular death
nonfatal myocardial infarction | 12 months
  Occurrence of nonfatal myocardial infarction
nonfatal stroke | 12 months
  Occurrence of of nonfatal stroke
ischemia-driven revascularization | 12 months
  Occurrence of ischemia-driven revascularization
hospitalization for unstable angina | 12 months
  Occurrence of hospitalization for unstable angina
stent/scaffold thrombosis | 12 months
  Occurrence of stent/scaffold thrombosis
in-stent restenosis | 12 months
  Occurrence of in-stent restenosis
bleeding | 12 months
  Occurrence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Cheng, Doctor, Principal Investigator — Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No